CLINICAL TRIAL: NCT00529308
Title: Transcranial Magnetic Stimulation for Individuals With Tourette's Syndrome
Brief Title: Transcranial Magnetic Stimulation (TMS) for Individuals With Tourette's Syndrome
Acronym: TMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Tourette Association of America (Other)
Responsible Party: Principal Investigator, Angeli Landeros-Weisenberger, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5480
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Tourette Syndrome
Keywords: Tourette; Tourette's
MeSH Terms: conditions — Tourette Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation (active)
- Sham (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation (sham)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (active) — Magstim Rapid2 stimulator with Air Film Coil at 110% motor threshold at 1Hz for 30 minutes.
  Other Names: Magstim Rapid2
  Arms: Active
Device: Transcranial Magnetic Stimulation (sham) — Magstim Rapid2 stimulator with Sham Air Film Coil at 110% motor threshold at 1Hz for 30 minutes.
  Other Names: Magstim Rapid2
  Arms: Sham

SUMMARY:
This study will evaluate the clinical efficacy of 1 Hz repetitive transcranial magnetic stimulation (rTMS) applied to the supplementary motor area (SMA) in Tourette's Syndrome (TS) patients who have not fully responded to conventional therapies. The investigators will collect TMS measures of motor cortex excitability to test whether rTMS restores normal levels of intracortical inhibition found to be deficient in TS. The investigators will administer neuropsychological tests to demonstrate that SMA targeted rTMS can be administered safely without significant impairments of cognitive or motor functioning. The investigators hypothesize that:

1. Compared to sham (placebo), active rTMS will improve symptoms of TS as assessed with the Yale Global Tic Severity Scale (Y-GTSS) and Clinical Global Impression (CGI).
2. Active (but not sham) rTMS will normalize levels of motor cortex excitability, as reflected by increased intracortical inhibition, motor threshold, and cortical silent period, and by decreased intracortical facilitation, relative to pre-treatment baseline.

DETAILED DESCRIPTION:
This study tests the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) in the treatment of Tourette's Syndrome (TS). It also examines measures of brain function to study the brain basis underlying TS.

Despite major advances in the study and treatment of TS, patients often do not experience full remission from pharmacotherapy or behavioral therapy (Leckman 2002). rTMS is a non-invasive procedure that stimulates the brain using magnetic fields. This pilot study reported that rTMS may reduce TS symptoms (Mantovani et al., 2006). While promising, prior research has several limitations (e.g., relatively small sample sizes, and lack of sham [placebo] comparison).

This study addresses the drawbacks of prior work, and will provide data that will help to determine whether rTMS can be useful for TS patients resistant to conventional therapies. 25 outpatients with TS who have been only partially responsive to conventional therapies will be randomly assigned to either active low frequency (1 Hz) rTMS or sham (placebo) stimulation. The active or sham stimulation will be applied to the supplementary motor area (SMA) daily for three weeks. If rTMS will be added onto ongoing pharmacotherapy, the doses must have been stable for four weeks prior to study entry. The SMA was selected because of its connections with brain areas implicated in TS. Pilot work indicates that stimulation of SMA with low frequency rTMS is beneficial in TS patients. Low frequency rTMS has the added benefit of a better safety profile (i.e. no risk of seizure) than high frequency rTMS.

Rating scales for symptom change will be obtained at baseline, during the rTMS course, and at the end of three weeks of treatment. Patients will then be offered an open-label cross-over phase for an additional three weeks of daily active rTMS treatment. Patients who meet remission criteria in either phase or response criteria following the cross-over phase will continue routine clinical care under the supervision of their treating psychiatrist and will be invited back for assessment at 1, 3, and 6 months to determine the persistence of benefit.

Excitability of the motor cortex has been reported to be abnormal in TS, and may relate to dysfunction in motor pathways. We will collect measures of motor cortex excitability (with single and paired-pulse TMS) at baseline and after each phase to study whether changes in these measures may be correlated with clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Tourette's Syndrome, as confirmed by the DSM-IV-TR criteria
* Residual TS symptoms, defined as a total Y-GTSS total motor tic or phonic tic score > 20, despite treatment with an adequate trial of medications (defined as a failure to respond to a trial of commonly used medications for TS such as clonidine, guanfacine, or neuroleptic medications, given at recommended dosage and duration based on the clinician's judgment)
* Persistent high level of tic severity for 4 months despite efforts to control the tics using medications, or the presence of self injurious tics
* Duration of the index episode of at least a year
* Individuals who cannot tolerate medications of class and dose at the specified duration as described above will also be included
* Patients currently on medication must be at the same stable dose(s) for one month prior to enrollment and be willing to continue at the same dose(s) through the duration of the study

Exclusion Criteria:

* Individuals diagnosed with major depressive disorder (current) of moderate or severe intensity (CGI ≥ 4), bipolar disorder (lifetime), any psychotic disorder (lifetime), or an Axis II personality disorder; with a history of substance abuse or dependence within the past year (except nicotine and caffeine); or at significant acute suicide risk will be excluded

Other exclusion criteria include those common to every TMS protocol:

* Individuals with a clinically defined neurological disorder, with an increased risk of seizure for any reason, with a history of treatment with TMS, deep brain stimulation for any disorder will be excluded
* Patients with cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed will be excluded
* Current use of any investigational drug, any medications with proconvulsive action, such as bupropion, maprotiline, tricyclic antidepressant, clomipramine, classical antipsychotics, and daily use of any medications with a known inhibitory effect on cortical excitability measures (e.g., anticonvulsants, standing doses of benzodiazepines, sedative/hypnotics, and atypical antipsychotics) will not be permitted
* If participating in psychotherapy, patients must have been in stable treatment for at least three months prior to entry into the study, with no anticipation of change in frequency therapeutic sessions, or the therapeutic focus over the duration of the TMS trial
* Finally, current significant laboratory abnormality, known or suspected pregnancy, women who are breast-feeding or women of childbearing potential not using a medically accepted form of contraception when engaging in sexual intercourse will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Mantovani, MD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Background] Alexander GE, Crutcher MD, DeLong MR. Basal ganglia-thalamocortical circuits: parallel substrates for motor, oculomotor, "prefrontal" and "limbic" functions. Prog Brain Res. 1990;85:119-46. PMID 2094891
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Artola A, Brocher S, Singer W. Different voltage-dependent thresholds for inducing long-term depression and long-term potentiation in slices of rat visual cortex. Nature. 1990 Sep 6;347(6288):69-72. doi: 10.1038/347069a0. PMID 1975639
- [Background] Bliss TV, Gardner-Medwin AR. Long-lasting potentiation of synaptic transmission in the dentate area of the unanaestetized rabbit following stimulation of the perforant path. J Physiol. 1973 Jul;232(2):357-74. doi: 10.1113/jphysiol.1973.sp010274. PMID 4727085
- [Background] Bruggeman R, van der Linden C, Buitelaar JK, Gericke GS, Hawkridge SM, Temlett JA. Risperidone versus pimozide in Tourette's disorder: a comparative double-blind parallel-group study. J Clin Psychiatry. 2001 Jan;62(1):50-6. doi: 10.4088/jcp.v62n0111. PMID 11235929
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Elwood RW. The California Verbal Learning Test: psychometric characteristics and clinical application. Neuropsychol Rev. 1995 Sep;5(3):173-201. doi: 10.1007/BF02214761. PMID 8653108
- [Background] Greenberg BD, Ziemann U, Cora-Locatelli G, Harmon A, Murphy DL, Keel JC, Wassermann EM. Altered cortical excitability in obsessive-compulsive disorder. Neurology. 2000 Jan 11;54(1):142-7. doi: 10.1212/wnl.54.1.142. PMID 10636140
- [Background] Hoffman RE, Cavus I. Slow transcranial magnetic stimulation, long-term depotentiation, and brain hyperexcitability disorders. Am J Psychiatry. 2002 Jul;159(7):1093-102. doi: 10.1176/appi.ajp.159.7.1093. PMID 12091184
- [Background] Kirkwood A, Dudek SM, Gold JT, Aizenman CD, Bear MF. Common forms of synaptic plasticity in the hippocampus and neocortex in vitro. Science. 1993 Jun 4;260(5113):1518-21. doi: 10.1126/science.8502997.
- [Background] Leckman JF. Tourette's syndrome. Lancet. 2002 Nov 16;360(9345):1577-86. doi: 10.1016/S0140-6736(02)11526-1. PMID 12443611
- [Background] Leckman JF, Hardin MT, Riddle MA, Stevenson J, Ort SI, Cohen DJ. Clonidine treatment of Gilles de la Tourette's syndrome. Arch Gen Psychiatry. 1991 Apr;48(4):324-8. doi: 10.1001/archpsyc.1991.01810280040006. PMID 2009034
- [Background] Leckman JF, Vaccarino FM, Kalanithi PS, Rothenberger A. Annotation: Tourette syndrome: a relentless drumbeat--driven by misguided brain oscillations. J Child Psychol Psychiatry. 2006 Jun;47(6):537-50. doi: 10.1111/j.1469-7610.2006.01620.x. PMID 16712630
- [Background] Marsh R, Alexander GM, Packard MG, Zhu H, Wingard JC, Quackenbush G, Peterson BS. Habit learning in Tourette syndrome: a translational neuroscience approach to a developmental psychopathology. Arch Gen Psychiatry. 2004 Dec;61(12):1259-68. doi: 10.1001/archpsyc.61.12.1259. PMID 15583117
- [Background] Moll GH, Heinrich H, Gevensleben H, Rothenberger A. Tic distribution and inhibitory processes in the sensorimotor circuit during adolescence: a cross-sectional TMS study. Neurosci Lett. 2006 Jul 31;403(1-2):96-9. doi: 10.1016/j.neulet.2006.04.021. Epub 2006 May 9. PMID 16690208
- [Background] Peterson BS, Leckman JF. The temporal dynamics of tics in Gilles de la Tourette syndrome. Biol Psychiatry. 1998 Dec 15;44(12):1337-48. doi: 10.1016/s0006-3223(98)00176-0. PMID 9861477
- [Background] Peterson BS, Skudlarski P, Anderson AW, Zhang H, Gatenby JC, Lacadie CM, Leckman JF, Gore JC. A functional magnetic resonance imaging study of tic suppression in Tourette syndrome. Arch Gen Psychiatry. 1998 Apr;55(4):326-33. doi: 10.1001/archpsyc.55.4.326. PMID 9554428
- [Background] Peterson BS, Staib L, Scahill L, Zhang H, Anderson C, Leckman JF, Cohen DJ, Gore JC, Albert J, Webster R. Regional brain and ventricular volumes in Tourette syndrome. Arch Gen Psychiatry. 2001 May;58(5):427-40. doi: 10.1001/archpsyc.58.5.427. PMID 11343521
- [Background] Peterson BS, Thomas P, Kane MJ, Scahill L, Zhang H, Bronen R, King RA, Leckman JF, Staib L. Basal Ganglia volumes in patients with Gilles de la Tourette syndrome. Arch Gen Psychiatry. 2003 Apr;60(4):415-24. doi: 10.1001/archpsyc.60.4.415. PMID 12695320
- [Background] Piacentini J, Chang S. Behavioral treatments for Tourette syndrome and tic disorders: state of the art. Adv Neurol. 2001;85:319-31. No abstract available. PMID 11530440
- [Background] Quintana H. Transcranial magnetic stimulation in persons younger than the age of 18. J ECT. 2005 Jun;21(2):88-95. doi: 10.1097/01.yct.0000162556.02720.58. PMID 15905749
- [Background] Rossi S, Pasqualetti P, Rossini PM, Feige B, Ulivelli M, Glocker FX, Battistini N, Lucking CH, Kristeva-Feige R. Effects of repetitive transcranial magnetic stimulation on movement-related cortical activity in humans. Cereb Cortex. 2000 Aug;10(8):802-8. doi: 10.1093/cercor/10.8.802. PMID 10920051
- [Background] Sallee FR, Kurlan R, Goetz CG, Singer H, Scahill L, Law G, Dittman VM, Chappell PB. Ziprasidone treatment of children and adolescents with Tourette's syndrome: a pilot study. J Am Acad Child Adolesc Psychiatry. 2000 Mar;39(3):292-9. doi: 10.1097/00004583-200003000-00010. PMID 10714048
- [Background] Sallee FR, Nesbitt L, Jackson C, Sine L, Sethuraman G. Relative efficacy of haloperidol and pimozide in children and adolescents with Tourette's disorder. Am J Psychiatry. 1997 Aug;154(8):1057-62. doi: 10.1176/ajp.154.8.1057. PMID 9247389
- [Background] Scahill L, Chappell PB, Kim YS, Schultz RT, Katsovich L, Shepherd E, Arnsten AF, Cohen DJ, Leckman JF. A placebo-controlled study of guanfacine in the treatment of children with tic disorders and attention deficit hyperactivity disorder. Am J Psychiatry. 2001 Jul;158(7):1067-74. doi: 10.1176/appi.ajp.158.7.1067. PMID 11431228
- [Background] Scahill L, Leckman JF, Schultz RT, Katsovich L, Peterson BS. A placebo-controlled trial of risperidone in Tourette syndrome. Neurology. 2003 Apr 8;60(7):1130-5. doi: 10.1212/01.wnl.0000055434.39968.67. PMID 12682319
- [Background] Scahill L, Riddle MA, King RA, Hardin MT, Rasmusson A, Makuch RW, Leckman JF. Fluoxetine has no marked effect on tic symptoms in patients with Tourette's syndrome: a double-blind placebo-controlled study. J Child Adolesc Psychopharmacol. 1997 Summer;7(2):75-85. doi: 10.1089/cap.1997.7.75. PMID 9334893
- [Background] Schultz RT, Carter AS, Gladstone M, Scahill L, Leckman JF, Peterson BS, Zhang H, Cohen DJ, Pauls D. Visual-motor integration functioning in children with Tourette syndrome. Neuropsychology. 1998 Jan;12(1):134-145. doi: 10.1037//0894-4105.12.1.134. PMID 9460741
- [Background] Shapiro E, Shapiro AK, Fulop G, Hubbard M, Mandeli J, Nordlie J, Phillips RA. Controlled study of haloperidol, pimozide and placebo for the treatment of Gilles de la Tourette's syndrome. Arch Gen Psychiatry. 1989 Aug;46(8):722-30. doi: 10.1001/archpsyc.1989.01810080052006. PMID 2665687
- [Background] Speer AM, Willis MW, Herscovitch P, Daube-Witherspoon M, Shelton JR, Benson BE, Post RM, Wassermann EM. Intensity-dependent regional cerebral blood flow during 1-Hz repetitive transcranial magnetic stimulation (rTMS) in healthy volunteers studied with H215O positron emission tomography: II. Effects of prefrontal cortex rTMS. Biol Psychiatry. 2003 Oct 15;54(8):826-32. doi: 10.1016/s0006-3223(03)00324-x. PMID 14550682
- [Background] Stanton PK, Sejnowski TJ. Associative long-term depression in the hippocampus induced by hebbian covariance. Nature. 1989 May 18;339(6221):215-8. doi: 10.1038/339215a0. PMID 2716848
- [Background] Wirshing DA, Boyd JA, Meng LR, Ballon JS, Marder SR, Wirshing WC. The effects of novel antipsychotics on glucose and lipid levels. J Clin Psychiatry. 2002 Oct;63(10):856-65. doi: 10.4088/jcp.v63n1002. PMID 12416594
- [Background] Ziemann U, Paulus W, Rothenberger A. Decreased motor inhibition in Tourette's disorder: evidence from transcranial magnetic stimulation. Am J Psychiatry. 1997 Sep;154(9):1277-84. doi: 10.1176/ajp.154.9.1277. PMID 9286189
- [Background] Parent A, Hazrati LN. Functional anatomy of the basal ganglia. I. The cortico-basal ganglia-thalamo-cortical loop. Brain Res Brain Res Rev. 1995 Jan;20(1):91-127. doi: 10.1016/0165-0173(94)00007-c. PMID 7711769
- [Background] Cohen LG, Roth BJ, Nilsson J, Dang N, Panizza M, Bandinelli S, Friauf W, Hallett M. Effects of coil design on delivery of focal magnetic stimulation. Technical considerations. Electroencephalogr Clin Neurophysiol. 1990 Apr;75(4):350-7. doi: 10.1016/0013-4694(90)90113-x. PMID 1691084
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Orth M, Kirby R, Richardson MP, Snijders AH, Rothwell JC, Trimble MR, Robertson MM, Munchau A. Subthreshold rTMS over pre-motor cortex has no effect on tics in patients with Gilles de la Tourette syndrome. Clin Neurophysiol. 2005 Apr;116(4):764-8. doi: 10.1016/j.clinph.2004.10.003. Epub 2004 Nov 25. PMID 15792884
- [Background] Wilhelm S, Deckersbach T, Coffey BJ, Bohne A, Peterson AL, Baer L. Habit reversal versus supportive psychotherapy for Tourette's disorder: a randomized controlled trial. Am J Psychiatry. 2003 Jun;160(6):1175-7. doi: 10.1176/appi.ajp.160.6.1175. PMID 12777279
- [Background] Bloch MH, Leckman JF, Zhu H, Peterson BS. Caudate volumes in childhood predict symptom severity in adults with Tourette syndrome. Neurology. 2005 Oct 25;65(8):1253-8. doi: 10.1212/01.wnl.0000180957.98702.69. PMID 16247053
- [Background] Chae JH, Nahas Z, Wassermann E, Li X, Sethuraman G, Gilbert D, Sallee FR, George MS. A pilot safety study of repetitive transcranial magnetic stimulation (rTMS) in Tourette's syndrome. Cogn Behav Neurol. 2004 Jun;17(2):109-17. doi: 10.1097/01.wnn.0000116253.78804.3a. PMID 15453520
- [Background] Davis KK, Davis JS, Dowler L. In motion, out of place: the public space(s) of Tourette Syndrome. Soc Sci Med. 2004 Jul;59(1):103-12. doi: 10.1016/j.socscimed.2003.10.008. PMID 15087147
- [Background] Fried I, Katz A, McCarthy G, Sass KJ, Williamson P, Spencer SS, Spencer DD. Functional organization of human supplementary motor cortex studied by electrical stimulation. J Neurosci. 1991 Nov;11(11):3656-66. doi: 10.1523/JNEUROSCI.11-11-03656.1991. PMID 1941101
- [Background] Karadenizli D, Dilbaz N, Bayam G. Gilles de la Tourette syndrome: response to electroconvulsive therapy. J ECT. 2005 Dec;21(4):246-8. doi: 10.1097/01.yct.0000184618.00661.72. PMID 16301887
- [Background] Knowlton BJ, Mangels JA, Squire LR. A neostriatal habit learning system in humans. Science. 1996 Sep 6;273(5280):1399-402. doi: 10.1126/science.273.5280.1399. PMID 8703077
- [Background] Mantovani A, Lisanby SH, Pieraccini F, Ulivelli M, Castrogiovanni P, Rossi S. Repetitive transcranial magnetic stimulation (rTMS) in the treatment of obsessive-compulsive disorder (OCD) and Tourette's syndrome (TS). Int J Neuropsychopharmacol. 2006 Feb;9(1):95-100. doi: 10.1017/S1461145705005729. Epub 2005 Jun 28. PMID 15982444
- [Background] Munchau A, Bloem BR, Thilo KV, Trimble MR, Rothwell JC, Robertson MM. Repetitive transcranial magnetic stimulation for Tourette syndrome. Neurology. 2002 Dec 10;59(11):1789-91. doi: 10.1212/01.wnl.0000036615.25044.50. PMID 12473773
- [Derived] Landeros-Weisenberger A, Mantovani A, Motlagh MG, de Alvarenga PG, Katsovich L, Leckman JF, Lisanby SH. Randomized Sham Controlled Double-blind Trial of Repetitive Transcranial Magnetic Stimulation for Adults With Severe Tourette Syndrome. Brain Stimul. 2015 May-Jun;8(3):574-81. doi: 10.1016/j.brs.2014.11.015. Epub 2014 Dec 3. PMID 25912296
- See also: Study summary on Brain Stimulation Division web site — http://www.brainstimulation.columbia.edu/research/clinical/tourette.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS | Sham
Started | 9 | 11
Completed | 8 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active: Magstim Rapid2 stimulator with Air Film Coil at 110% motor threshold at 1Hz for 30 minutes.
- Sham: Magstim Rapid2 stimulator with Sham Air Film Coil at 110% motor threshold at 1Hz for 30 minutes.
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (7.4) | 39.0 (16.1) | 33.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Yale Global Tic Severity Scale (Y-GTSS)
Description: Y-GTSS is a clinician-rated scale used to assess tic severity. Motor and phonic tics are rated separately from 0 to 5 on several scales including number, frequency, intensity, complexity, and interference. Thus Motor and Phonic Tic scores can range from 0 to 25; the combined Total Tic Score ranges from 0 to 50. There is also an Impairment score that rates the overall burden due to tics. The Impairment scale yields a single score from 0 to 50 with higher scores indicating higher levels of overall impairment associated with tics.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 9 | 11
units on a scale | 29.5 (11.9) | 31.5 (8.1)

2. Primary Outcome: Motor Cortex Excitability Normalization-Right Motor Threshold
Description: Motor Threshold (MT) is thought to be a measure of membrane excitability in pyramidal neurons. MT is defined as the minimum magnetic flux needed to elicit a threshold EMG response (50 µV in peak to peak amplitude) in a resting target muscle in 5 out of 10 trials using single pulse TMS administered to the contralateral primary motor cortex. MT for both right and left hand are determined, and the lowest is used to select the intensity for rTMS.
Time Frame: 3 weeks
Population: This data was only available for the subjects at the Yale site only.
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Active | Sham
Number analyzed (Participants) | 4 | 9
µV | 56 (16.3) | 59.8 (16.3)

3. Primary Outcome: Number of Patients With "Much Improved or Very Much Improved" on Clinical Global Impression-Improvement (CGI) Scale
Description: The CGI-I is a clinician-rated scales that have been used in clinical trials for over 25 years. Clinicians rate patient improvement compared to baseline. By convention, 4 = No Change; scores of 5, 6, and 7 move in the direction of worsening; scores of 3, 2, and 1 correspond to "Minimal Improvement," "Much Improved" or "Very Much Improved," respectively. CGI-I ratings of "Much" or "Very Much Improved" at post-treatment are used to identify treatment responders.
Time Frame: 3 weeks
Measure: Number; unit: participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 9 | 11
participants | 1 | 0

4. Primary Outcome: Motor Cortex Excitability Normalization-Left Motor Threshold
Description: as for outcome 2
Time Frame: 3 weeks
Population: This data was only available for the subjects at the Yale site only.
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Active | Sham
Number analyzed (Participants) | 4 | 9
µV | 56.5 (12.8) | 63.8 (16.3)

5. Primary Outcome: Number of Patients With "Improved or Minimally Improved" in Clinical Global Impression-Improvement (CGI) Scale
Description: as for outcome 3
Time Frame: 3 weeks
Measure: Number; unit: participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 9 | 11
participants | 2 | 8

ADVERSE EVENTS:
Time Frame: Adverse Events were collected throughout the duration of the study, which was approximately 4 years.
Arm/Group | Active | Sham
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 4/8 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=8) | Sham (N=10)
Headache (Nervous system disorders) | 4 | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 9
Scalp Pain (Skin and subcutaneous tissue disorders) | 2 | 2
Trouble Concentrating (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes